CLINICAL TRIAL: NCT04006769
Title: Entacapone in Combination With Imatinib Mesylate for Treatment of Patients With Gastrointestinal Stromal Tumors(GIST) Following Failure of at Least Imatinib and Sunitinib
Brief Title: Entacapone Combination With Imatinib for Treatment of GIST
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Lun-Quan Sun, Director of Center for molecular medicine, Xiangya hospital, Central South University, Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gist-ent
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Stromal Tumor, Malignant
Keywords: entacapone; Imatinib mesylate; GIST; treatment
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — entacapone; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Entacapone & Imatinib mesylate (Experimental): Entacapone 200mg tablet (Orion pharma,Switzerland) by mouth, three times a day and then escalated to final dose of 1.0 grams three times per day within one week, until disease progression, intolerable toxicity, or withdrawal of informed consent, whichever occurs first.
  And Imatinib mesylate 400mg tablet by mouth, once a day until disease progression, intolerable toxicity, or withdrawal of informed consent, whichever occurs first.
  Interventions: Drug: Entacapone; Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Entacapone — Entacapone tablet
  Other Names: Comtan; Comtess
Drug: Imatinib Mesylate — Imatinib Mesylate tablet
  Other Names: Gleevec

SUMMARY:
This study evaluates the combination of entacapone and imatinib in the treatment of gastrointestinal stromal Tumors who have progressed on the setting of at least Imatinib and Sunitinib. 5 participants will be included in this open-label observatory study.

DETAILED DESCRIPTION:
The eligibility criteria are patients whose histologically confirmed disease which is currently metastatic/unresectable gastrointestinal stroma tumor (GIST) of c-KIT E11 mutation genotype. He received imatinib as the first-line treatment and no progression within the first 6 months (no primary resistance to imatinib), with disease progression following treatment with at least imatinib and sunitinib, and at least 1 measurable lesion (the longest diameter≥ 10mm). Age should be more or equal 18 years with adequate hematologic and end-organ function and good performance ((ECOG PS) ≤ 2, or 3 (the symptoms were definitely caused by GIST itself).

This study is single group assignment and open label. The intervention/treatment is Entacapone combined with Imatinib. Entacapone began with 200mg tablet (Orion pharma, Switzerland) by mouth, three times a day and then escalated to final dose of 1.0 grams three times per day within one week, until disease progression, intolerable toxicity, or withdrawal of informed consent, whichever occurs first. Imatinib mesylate 400mg tablet by mouth, once a day until disease progression, intolerable toxicity, or withdrawal of informed consent, whichever occurs first. Periodically routine blood test including liver and kidney function, troponin and electrocardiogram were conducted throughout the entire clinical course.

Clinic visits are performed at 16 points: visit 1, baseline, and then follow up after first dose as planned: 1st month, and every 2 months in the first year, followed by every 3 months until 3 years or 31 days after withdraw. The study design is visualized in Figure 1 below.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and comply with the requirements of the study and the schedule of assessments.
2. Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
3. Expected life span > 12 weeks.
4. Histologically confirmed disease which is currently metastatic/unresectable gastrointestinal stroma tumor(GIST) of c-KIT E11 mutation genotype.
5. Patients received imatinib as the first-line treatment and no progression within the first 6 months(no primary resistance to imatinib ). With disease progression following treatment with at least imatinib and sunitinib.
6. Patients must be able to provide archival tumor tissues (approximately 4 [at least 2] unstained Formalin Fixed and Paraffin Embedded Tissues （FFPET）slides) for biomarker analysis to assess the expression of FTO and c-KIT protein.
7. At least 1 measurable lesion (the longest diameter≥ 10mm). Note: Computed Tomography（CT） abdomen and pelvis with contrast including peritoneum, or positron emission tomography/computed tomography(PET/CT) performed skull base to knees or whole body before the first day of entacapone.
8. Eastern Cooperative Oncology Group-performance status(ECOG PS) ≤ 2,or 3(the symptoms were definitely caused by GIST itself).
9. Adequate hematologic and end-organ function, as defined by the following laboratory results (obtained ≤ 28 days prior to the first day of entacapone):

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10 9 /L, hemoglobin ≥ 80 g/L and platelets ≥80 × 10 9 /L.
   * Total serum bilirubin ≤ 2.5 × upper limit of normal (ULN); Aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5× ULN.
   * Estimated creatinine clearance rate≥ 60 mL/min（According to the formula of Cockcroft-Gault）.
10. Females of childbearing potential must be willing to practice highly effective method of birth control for the duration of the study, and at least 120 days after the last dose of entacapone or imatinib. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and at least 120 days after the last dose of entacapone or imatinib.

Exclusion Criteria:

1. Age < 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
2. Progression within the first 6 months of first-line imatinib treatment (primary imatinib resistance).
3. Patients with active/symptomatic carrier or chronic hepatitis B virus (HBV) whose HBV DNA ≥ 1×104 copies/mL should be excluded. Note: Patients with detectable hepatitis B surface antigen(HBsAg) or HBV DNA should be managed per treatment guidelines. Patients receiving antivirals at screening should have been treated for ≥2 weeks prior to written informed consent and should continue treatment for 6 months after study drug treatment discontinues.

   Note: Patients with active hepatitis C may enroll and those with detectable hepatitis C virus(HCV) RNA who are receiving antiviral therapy at time of screening should remain on continuous, effective antiviral therapy during the study.
4. A known history of human immunodeficiency virus(HIV) infection.
5. Malignancy other than GIST and still under the active treatment.
6. Was administered a live vaccine ≤ 4 weeks before written informed consent.
7. Any of the following medical conditions may threaten the safety of patients or affect the trial obedience including symptomatic heart failure requiring systematic treatment, unstable angina , acute myocardial infarction and severe chronic or active infections (including tuberculosis infection) requiring systemic antibacterial, antifungal, or antiviral therapy.
8. History of severe hypersensitivity reactions to any ingredient of entacapone and imatinib.
9. Pheochromocytoma or history of neuroleptic malignant syndrome(NMS) and/or non-traumatic rhabdomyolysis (NRML).
10. Female in pregnancy or lactation(Urine or serum pregnancy test and documented as negative within 7 days prior to the first dose of entacapone for the female with fertility expectation or sexual intercourse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) And Serious Adverse Events(SAE) | 36 months or 31 days after last dose, which come first.
  According to Criteria CTCAE5.0, the ratio of AE and SAE which were defined by the Common Terminology Criteria for Adverse Events, CTCAE.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 36 Months
  The ORR is the proportion of the patients who achieved complete response (CR) or partial responses(PR) according to CHOI criteria.
Quality of Life(QOL) | Difference between baseline and the timepoint of the best efficacy within 181 days.
  The data was collected using EORTC QLQ-C30 V3.0 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bin Li, MD, Principal Investigator — Xiangya Hospital, Central South University, Changsha, Hunan,China,410008
Locations (1):
- Bin Li, MD, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting at the 6 months after publication.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Background] Tabone S, Theou N, Wozniak A, Saffroy R, Deville L, Julie C, Callard P, Lavergne-Slove A, Debiec-Rychter M, Lemoine A, Emile JF. KIT overexpression and amplification in gastrointestinal stromal tumors (GISTs). Biochim Biophys Acta. 2005 Jun 30;1741(1-2):165-72. doi: 10.1016/j.bbadis.2005.03.011. Epub 2005 Apr 13. PMID 15869870
- [Background] Peng S, Xiao W, Ju D, Sun B, Hou N, Liu Q, Wang Y, Zhao H, Gao C, Zhang S, Cao R, Li P, Huang H, Ma Y, Wang Y, Lai W, Ma Z, Zhang W, Huang S, Wang H, Zhang Z, Zhao L, Cai T, Zhao YL, Wang F, Nie Y, Zhi G, Yang YG, Zhang EE, Huang N. Identification of entacapone as a chemical inhibitor of FTO mediating metabolic regulation through FOXO1. Sci Transl Med. 2019 Apr 17;11(488):eaau7116. doi: 10.1126/scitranslmed.aau7116. PMID 30996080
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774